CLINICAL TRIAL: NCT02856243
Title: Direct Antiviral Agents for Hepatitis C Virus-associated Cryoglobulinaemia Vasculitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: VASCUVALDIC 2 study
Record Dates: First submitted 2016-07-19; First posted 2016-08-04 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-07

CONDITIONS: Vasculitis; Cryoglobulinemia; Hepatitis C
MeSH Terms: conditions — Vasculitis; Cryoglobulinemia; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: new antiviral therapy

SUMMARY:
Cryoglobulinemia are responsible for systemic vasculitis, and the most frequently targeted organs are the skin, joints, kidney and peripheral nervous system. Cryoglobulinemia vasculitides are associated with significant morbidity and mortality, and require therapeutic intervention. With the discovery of hepatitis C virus (HCV) as the etiologic agent for most cases of mixed cryoglobulinemia new opportunities and problems for crafting therapy of HCV mixed cryoglobulinemia (MC) have emerged. A new and major concern was the potential adverse effects that immunosuppressive therapy with glucocorticoids and cytotoxic drugs could have on an underlying chronic viral infection. Alternatively the discovery of HCV provided the opportunity to control HCV-MC with antiviral therapy based on the belief that the underlying infection was driving immune complex formation and resultant vasculitis. Inducing a sustained virologic and clinical response and minimizing the use of immunosuppressive drugs are the main goals in the treatment of patients with HCV-MC vasculitis. Aggressive antiviral therapy has been shown to induce a complete remission of HCV-MC in up to 70% of patients. New antiviral combination, Interferon (IFN)-free regimens have recently proved very high virological response rate and with a very good safety profile and now need to be evaluated in severe and/or refractory HCV-MC patient's population.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age or older
* present an active HCV vasculitis defined by a clinically active vasculitis with skin, joint, renal, peripheral nerve, central neurological, digestive, pulmonary and/or cardiac involvement (no histological evidence needed if patient had purpura)
* chronic active HCV infection (positive HCV RNA)
* informed consent

Exclusion Criteria:

* non-active cryoglobulinaemia vasculitis
* HIV
* active hepatitis B virus (HBV) infection
* current decompensated cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be eligible, the patient must have been at least 18 years of age or older, without any upper age limit, informed and present an active HCV vasculitis defined by a clinically active vasculitis with skin, joint, renal, peripheral nerve, central neurological, digestive, pulmonary and/or cardiac involvement (no histological evidence needed if patient had purpura), and a chronic active HCV infection (positive HCV RNA).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete clinical response of cryoglobulinaemia vasculitis | At week 24
  The complete clinical response is defined by improvement of all the affected organs involved at baseline and the absence of clinical relapse. The skin and articular improvement will be evaluated clinically (i.e. disappearance of purpura and/or ulcers and/or skin necrosis, disappearance of arthralgia and/or arthritis). Renal improvement will be evaluated biologically (i.e. proteinuria <0.3g/24h, disappearance of hematuria and improvement of Glomerular filtration rate (GFR) > 20% at week 24 if GFR < 60 ml/min/1.73 m² at diagnosis). Peripheral neurological improvement will be evaluated clinically (i.e. improvement of pains and paraesthesia by visual analogue scales, improvement of muscular testing in case of motor impairment at baseline) and/or electrophysiologically (i.e. improvement of electromyogram abnormalities at week 24 compared to baseline). The neuropathy total symptom score-6 (NTSS-6) will be applied to evaluate individual neuropathy sensory symptoms.

SECONDARY OUTCOMES:
Number of participants with sustained virological response | At week 36
  A sustained virological response is defined by the absence of detectable serum HCV RNA twelve weeks after the end of antiviral therapy
Number of participants with Immunological complete response | At week 36
  Immunological complete response is defined by negativation of cryoglobulin at week 36.
rate of side effects | up to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- hopital La pitié Salpétrière, Paris, France